CLINICAL TRIAL: NCT07104825
Title: Autonomic Neural Blockade During Sleeve Gastrectomy and Gastric Bypass: A Randomized Controlled Trial Evaluating Pain and Nausea After Bariatric Surgery
Brief Title: Autonomic Neural Blockade in Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Herbert Hedberg, Gastrointestinal and General Surgery Physician, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000229
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Bariatric Surgery Candidate; Pain, Postoperative; Nausea and Vomiting, Postoperative; Opioid Use
Keywords: Autonomic, blockade, bariatric surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: A single-blinded randomized controlled trial
Who Masked: Participant
Masking Description: The study participants will be blinded to treatment arm assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Paragastric Autonomic Neural Blockade (Experimental): ANB will be performed in addition to administration of local anesthetic to abdominal incisions (standard of care). The block is administered via syringe attached to IV tubing and 25g hypodermic needle. The needle and tubing are introduced through a laparoscopic port with the cap in place, and the needle is grasped and cap removed in the abdomen. The needle is advance into perigastric tissue along the lesser curve, the lack of vascular penetration is confirmed with aspiration, and the anesthetic (0.5% bupivacaine-10ml, 50mg and Liposomal bupivacaine-10ml, 133mg) is injected. 10ml is distributed along the lesser curve, and 5ml on either side of the celiac trunk, identified by dividing the lesser omentum and elevating the stomach.
  Interventions: Procedure: Intraoperative autonomic neural blockade (ANB)
- Laparoscopic Standard of Care Abdominal Wall Block (Active Comparator): Laparoscopic bariatric surgeries are performed with local anesthetic injected into the abdominal wall only. This may be with transversus abdominis block or local injection at the port sites. At our institution, standard of care is local injection at port sites with bupivacaine (30ml) spread among the five small incisions. This standard will be maintained for every patient in the study.
  Interventions: Procedure: Laparoscopic Standard of Care Abdominal Wall Block

INTERVENTIONS:
Procedure: Intraoperative autonomic neural blockade (ANB) — Local anesthetic block of the neurovascular tissue along the lesser curve of the stomach and celiac trunk during sleeve gastrectomy or gastric bypass surgery.
  Other Names: Neurovascular tissue block
  Arms: Laparoscopic Paragastric Autonomic Neural Blockade
Procedure: Laparoscopic Standard of Care Abdominal Wall Block — Administration of local anesthetic to abdominal incisions (standard of care)
  Other Names: Bariatric Surgery
  Arms: Laparoscopic Standard of Care Abdominal Wall Block

SUMMARY:
The purpose of this research is to evaluate if autonomic nerve block (ANB- blocking pain and nausea signals) decreases pain and anti-nausea medication requirements as well as the experience of pain/nausea during the first 72 hours after sleeve gastrectomy or gastric bypass surgery. Participants will be randomly assigned either to the standard of care or the ANB group before surgery. As part of standard of care, in both groups, laparoscopic bariatric surgery will be initiated with local anesthetic injected into the abdominal wall. In the ANB group, participants will be given an additional injection of local anesthetic medication to block nerves on and around the stomach.

DETAILED DESCRIPTION:
Gastric bypass and sleeve gastrectomy are the most common and successful weight loss surgeries. The advancement of laparoscopic, minimally invasive techniques allows these procedures to be performed with low morbidity and a relatively easy recovery, when broadly considering abdominal surgery. The major complaints postoperatively are abdominal pain and nausea, which can require medications to control and may prolong hospital stay. There is evidence autonomic neural blockade (ANB) improves pain and nausea in the immediate postoperative period. ANB has been shown to be therapeutic in the surgical environment providing extended analgesia for pain following surgery.

This study is a single-blinded randomized controlled trial comparing the total morphine milligram equivalents (MMEs) of pain medication used 72 hours post-operative period in patients who received the ANB vs standard of care. In the ANB group, additional local anesthetic block of the neurovascular tissue along the lesser curve of the stomach and celiac trunk will be performed using 0.5% bupivacaine 10ml, 50mg and Liposomal bupivacaine 10ml, 133mg dose. Study participants will not be told if they received the block, but the surgeon will be aware of which study group participants are assigned.

ELIGIBILITY:
Inclusion Criteria:

* Individuals able and willing to consent and participate in all study activities
* Adults, ages 18-90
* All patients with severe obesity undergoing laparoscopic/robotic gastric bypass or sleeve gastrectomy

Exclusion Criteria:

* Patients taking opiates chronically
* Patients allergic to study medications
* Patients with any prior adverse reaction to ingredients included in the block
* Adults unable to consent
* Pregnant women
* Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain medication consumed post-operatively | Post-op 72 hours
  Total Morphine milligram equivalents (MMEs) of pain medication utilized during the first 72hrs after bariatric surgery

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | Day of surgery, post-op days 1, 2 and 3.
  Numerical pain scale from 0 (no pain) to 10 (worst pain possible)
Nausea, retching and vomiting symptoms | Post-op days 1, 2 and 3.
  Proportion of patients reporting nausea, retching and vomiting on post-op days 1, 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hedberg, MD, Principal Investigator — Endeavor Health
Locations (1):
- Endeavor Health, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daes J, Pantoja R, Luque E, Hanssen A, Rocha J, Pauli EM. Intraoperative autonomic neural blockade: comparison between different local anesthetics combinations: a randomized clinical trial. Surg Endosc. 2025 Apr;39(4):2523-2533. doi: 10.1007/s00464-025-11637-0. Epub 2025 Mar 3. PMID 40032662
- [Background] Daes J, Pantoja R, Luquetta J, Luque E, Hanssen A, Rocha J, Morrell DJ. Impact on Anesthetic Agent Consumption After Autonomic Neural Blockade as Part of a Combined Anesthesia Protocol: A Randomized Clinical Trial. Anesth Analg. 2024 Sep 1;139(3):581-589. doi: 10.1213/ANE.0000000000006769. Epub 2023 Dec 13. PMID 38091501
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617